CLINICAL TRIAL: NCT06447636
Title: Perioperative Surufatinib Plus Sintilimab Combined With Chemotherapy in Locally Advanced Gastric and Gastroesophageal Junction Adenocarcinoma: the Phase 2 Solids-01 Trial
Brief Title: Perioperative Surufatinib Plus Sintilimab Combined With Chemotherapy in Gastric/Gastroesophageal Junction Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Fenglin Liu, MD PhD, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOLIDS-01
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Gastric Cancer; Gastro Esophageal Junction Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — surufatinib; sintilimab; Oxaliplatin; S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surufatinib，sintilimab and SOX chemotherapy (Experimental): Surufatinib: 250mg qd，d1-21, q3w; Surufatinib: 200mg, ivdrip, d1, q3w; SOX: Oxaliplatin+S-1 S-1:40~60mg Bid, d1~14, q3w; Oxaliplatin: 130mg/m2, ivdrip,d1, q3w; Neoadjuvant therapy for 2-4 cycles, adjuvant therapy for 3-5 cycles. After 6 cycles of SOX chemotherapy, Surufatinib + Surufatinib was taken orally until one year.
  Interventions: Drug: Surufatinib; Drug: Sintilimab; Drug: Oxaliplatin; Drug: S1

INTERVENTIONS:
Drug: Surufatinib — Surufatinib: 250mg qd，d1-21, q3w
Drug: Sintilimab — Sintilimab：200mg ivdrip, d1, q3w
Drug: Oxaliplatin — 130mg/m2，iv drip for 2h，d1, q3w
Drug: S1 — S1：40~60mg Bid，d1~14, q3w

SUMMARY:
For locally advanced gastric and gastroesophageal junction adenocarcinoma (cT3-4bNanyM0), perioperative PD-1 antibody combined with chemotherapy can downstage tumor stage, increase the R0 resection rate, and may improve the long-term survival. Combination of perioperative surufatinib, sintilimab and chemotherapy for locally advanced gastric and gastroesophageal junction adenocarcinoma could be a novel therapeutic strategy to increase response rate and therapeutic efficacy. Surufatinib, as the oral drug in this study is a small molecule kinase inhibitor that mainly acts on vascular growth factor receptor (VEGFR1, 2,3), fibroblast growth factor receptor 1(FGFR1) and colony stimulating factor 1 receptor (CSF1R). It is a proprietary product developed by Hutchison Whampoa Pharmaceutical (Shanghai, China) Co., LTD. Surufatinib has been approved for neuroendocrine tumor. This study is a monocenter, single-arm phase 2 clinical trial to evaluate tolerability, safety and efficacy of perioperative surufatinib in combination with sintilimab and chemotherapy in locally advanced gastric and gastroesophageal junction adenocarcinoma.

DETAILED DESCRIPTION:
The incidence of gastric and gastroesophageal junction adenocarcinoma is increasing in China, and it is one of the most common malignant tumors in China. Surgery is the only possible way to cure gastric and gastroesophageal junction adenocarcinoma, however, over 70-80% of gastric/gastroesophageal junction adenocarcinoma patients in China are in advanced stage. Locally gastric/gastroesophageal junction adenocarcinoma (cT3-4bNanyM0) could be cured by multi-disciplinary therapies including surgery, immunotherapy and chemotherapy. Perioperative immunotherapy plus chemotherapy can downstage tumor T and N stage, increase the R0 resection rate, and may improve the long-term survival. However, the therapeutic effects still not satisfactory to date. Surufatinib, as the novel oral antivascular targeting drug, has been proved to be effective in neuroendocrine tumor. Combination of perioperative surufatinib and immunotherapy plus chemotherapy for locally advanced gastric/gastroesophageal junction adenocarcinoma could be a novel therapeutic strategy to increase response rate and therapeutic efficacy. This study is a monocenter, single-arm phase 2 clinical trial to evaluate tolerability, safety and efficacy of perioperative surufatinib in combination with sintilimab and chemotherapy in locally advanced gastric and gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* patients age 18-75 years;
* Histologically CT/MRI confirmed cT3-4bNanyM0 gastric or GEJ adenocarcinoma;
* ECOG 0-1, no surgery contraindications;
* Expected survival ≥3 months;

Exclusion Criteria:

* signs of distant metastases
* Prior chemotherapy, radiotherapy, surgery for gastric cancer;
* Significant cardiovascular disease
* major surgical procedure within 4 weeks prior to initiation of study treatment
* current treatment with anti-viral therapy or HBV
* pregnancy or breastfeeding
* history of malignancy within 5 years prior to screening
* Present or history of any autoimmune disease or immune deficiency;
* Prior therapy with a PD-1, anti-PD-Ligand 1 (PD-L1) or CTLA-4 agent;
* There are active gastric and duodenal ulcers, ulcerative colitis and other gastrointestinal diseases, or active bleeding in unresectable tumors.
* Poorly controlled hypertension or diabetes;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response（pCR）rate | From the initiation date of first cycle (each cycle is 21 days) to the date of operation, an average of 12 weeks

SECONDARY OUTCOMES:
R0 resection rate | From the initiation date of first cycle (each cycle is 21 days) to the date of operation, an average of 12 weeks.
Disease free survival (DFS) | From the initiation date of first cycle (each cycle is 21 days) to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
Overall survival (OS) | From the initiation date of first cycle (each cycle is 21 days) to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No